CLINICAL TRIAL: NCT02539823
Title: To Characterize the Acute and Short-term Effects of Cannabidiol (CBD) Administration on Cue-induced Craving in Drug-abstinent Heroin-dependent Humans
Brief Title: Acute and Short-term Effects of CBD on Cue-induced Craving in Drug-abstinent Heroin-dependent Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hurd,Yasmin, Ph.D. (Individual)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Yasmin Hurd, Professor of Neuroscience, Psychiatry and Pharmacology & Systems Therapeutics, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSBI HSM# 087-14
Record Dates: First submitted 2015-08-25; First posted 2015-09-03 (Estimated); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Opiate Addiction
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): Subjects will receive a solution that resemble the Cannabidiol solution but do not have have its properties
  Interventions: Drug: Control (placebo)
- CBD 400mg (Experimental): Subjects will receive 400mg of cannabidiol
  Interventions: Drug: CBD 400 mg
- CBD 800mg (Experimental): Subjects will receive 800 mg of cannabidiol
  Interventions: Drug: CBD 800 mg

INTERVENTIONS:
Drug: CBD 400 mg — Subjects in Arm CBD 400 mg will receive 400mg of Cannabidiol in each of the three test sessions
  Other Names: CBD
  Arms: CBD 400mg
Drug: CBD 800 mg — Subjects in Arm CBD 800 mg will receive 800mg of Cannabidiol in each of the three test sessions
  Other Names: CBD
  Arms: CBD 800mg
Drug: Control (placebo) — Subjects will receive a harmless, inactive solution to compare and validate the results of the other arms of the study
  Other Names: CBD
  Arms: Control

SUMMARY:
Despite the current available therapies for opioid-dependent patients, most patients relapse. This research project focuses on the development of a novel compound, cannabidiol, to modulate opioid craving in humans based on animal models showing its selective effectiveness to inhibit drug-seeking behavior. The development of a targeted treatment for opioid relapse would be of tremendous medical and public health value.

DETAILED DESCRIPTION:
There has been an epidemic rise in heroin abuse and overdose in recent years. Of the more than one million people suffering today from opiate dependency, less than a quarter of such individuals receive treatment. Pharmacotherapeutic approaches traditionally have targeted mu opioid receptors since heroin and its metabolites bind with highest affinity to this receptor subtype. Although such treatment strategies have improved substance abuse outcomes, they do not effectively block opiate craving and thus are still associated with high rates of relapse. Using a strategy of indirectly regulating neural systems to modulate opioid-related behavior, our preclinical rodent studies consistently demonstrated that cannabidiol (CBD), a nonpsychoactive component of cannabis, specifically inhibited cue-induced heroin-seeking behavior. CBD's selective effect on drug-seeking behavior was pronounced after 24 hrs and endured even two weeks after the last drug administration following short-term CBD exposure. The fact that drug craving is generally triggered by exposure to conditioned cues suggests that CBD might be an effective treatment for heroin craving, specially given its protracted impact on behavior. CBD has already been shown in Phase I of our study and in various clinical studies to be well tolerated with a wide safety margin in human subjects. CBD thus represents a strong candidate for the development as a potential therapeutic agent in humans for opioid craving and relapse prevention. Preliminary pilot study showed CBD decreased craving. It is the goal of the current study to more fully characterize the effects of CBD administration on cue-induced craving in drug-abstinent heroin-dependent subjects using a random double blind design during a post-acute (greater than 6 days since last use) heroin withdrawal period. Study participants will be administered CBD during 3 test sessions and studied for the effects on cue-induced craving during those sessions as well as one week after the final CBD administration on the final test day (session 4).

ELIGIBILITY:
Inclusion Criteria:

* Must be between 21 and 65 years old
* Must have an opiate dependence that meets criteria set in the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM-V) Structured Clinical Interview for DSM (SCID-V) over the last three months
* No opioid use in the past 7 days (will be verified via urine drug screen and opiate metabolite test)

Exclusion Criteria:

* Using any psychoactive drug (other than nicotine) any time up to test session 3
* Having a diagnosis of drug dependence (except for heroin or nicotine) in the past 3 months, based on the SCID-V interview criteria
* Being maintained on methadone or buprenorphine, or taking opioid antagonists such as naltrexone
* Having a positive a drug screen
* Showing signs of acute heroin withdrawal symptoms
* Having medical conditions, including Axis I psychiatric conditions under DSM-V (examined using the Mini International Neuropsychiatric Interview [MINI])
* Having a a history of cardiac disease, arrhythmias, head trauma, and seizures
* Having a history of hypersensitivity to cannabinoids
* Arriving to the study site visibly intoxicated as determined by a clinical evaluation for signs and symptoms of intoxication and as verified by a drug screen
* Participating in a another pharmacotherapeutic trial in the past 3 months
* Being pregnant of breastfeeding
* Not using or irregularly using appropriate methods of contraception such as hormonal contraceptives (e.g., Depo-Provera, Nuva-Ring), an intrauterine device (IUD), or double barrier method (combination of any two barrier methods used simultaneously, e.g., condoms, spermicide, diaphragms)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Hurd, PhD, Principal Investigator — Mount Sinai Health System
Locations (1):
- Mount Sinai Beth Israel, New York, New York, United States

REFERENCES:
- [Derived] Hurd YL, Spriggs S, Alishayev J, Winkel G, Gurgov K, Kudrich C, Oprescu AM, Salsitz E. Cannabidiol for the Reduction of Cue-Induced Craving and Anxiety in Drug-Abstinent Individuals With Heroin Use Disorder: A Double-Blind Randomized Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):911-922. doi: 10.1176/appi.ajp.2019.18101191. Epub 2019 May 21. PMID 31109198

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | CBD 400mg | CBD 800mg
Started | 15 | 14 | 13
Completed | 15 | 14 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | CBD 400mg | CBD 800mg | Total
Number analyzed (Participants) | 15 | 14 | 13 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (8.0) | 51.9 (7.9) | 50.5 (11.6) | 49.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 12 | 12 | 11 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 1 | 1 | 5
  Black | 9 | 12 | 8 | 29
  Hispanic | 2 | 1 | 4 | 7
  Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 13 | 42

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cue-Induced In-Clinic Craving (From Baseline to Post-cue (30 Minutes), and From Test Day 1 Through Test Day 4 (1 Week)) - Via the Visual Analog Scale for Craving (VASC)
Description: The VASC will be administered to assess potential variations in the subjective craving effects associated with heroin. Following the administration of the investigational drug, craving induced in response to the cue sessions in the clinic will be measured. Note, cue sessions occur consecutively in the same test day. In this way, changes in craving from baseline (pre-cue to post-cue within each test day), as well as changes in cue-induced craving over the short-term (test day 1 through test day 4 a week later) will be monitored and measured. VASC scale ranges from 0 for "Not Craving at All" to 10 for "Extremely Craving."
Time Frame: VASC: test day I, II and IV - at arrival, baseline for cue 1 and 2, post-cue 1 and 2, before discharge (approximately 2.5 hours from session start on average); test day III: at arrival and discharge (approx. 2.5 hours from session start on average)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBD 400mg | CBD 800mg
Number analyzed (Participants) | 15 | 14 | 13
units on a scale
  First Baseline (before cue video) Session 1 | 1.40 (1.765) | 1.64 (1.946) | 2.31 (2.057)
  First Baseline (before cue video) Session 2 | 1.33 (1.33) | 1.07 (1.141) | 1.46 (2.106)
  First Baseline (before cue video) Session 4 | .53 (.53) | .79 (1.051) | 1.58 (2.429)
  First Post Cue Session 1 | 2.53 (3.091) | 2.21 (1.929) | 2.69 (1.932)
  First Post Cue Session 2 | 2.00 (2.646) | 1.36 (1.336) | 1.85 (2.512)
  First Post Cue Session 4 | 1.27 (1.710) | 1.07 (1.141) | 1.67 (2.498)
  Second Base Line (before cue video) Session 1 | 1.47 (2.326) | 1.43 (1.950) | 1.77 (1.878)
  Second Base Line (before cue video) Session 2 | 1.00 (1.363) | 1.00 (1.109) | 1.62 (2.022)
  Second Base Line (before cue video) Session 4 | .60 (1.121) | .79 (1.122) | 1.00 (1.595)
  Second Post Cue Session 1 | 2.40 (2.746) | 1.36 (1.598) | 1.69 (1.797)
  Second Post Cue Session 2 | 1.87 (2.696) | 1.79 (1.805) | 1.62 (2.219)
  Second Post Cue Session 4 | 1.20 (1.781) | .79 (1.188) | .75 (1.422)
  Post Relaxation video Session 1 | .33 (.617) | .93 (1.072) | 1.08 (1.188)
  Post Relaxation video Session 2 | .93 (1.280) | .64 (.842) | 1.00 (1.633)
  Post Relaxation video Session 4 | .33 (1.047) | .64 (1.008) | .58 (.900)

2. Primary Outcome: Changes in Out-of-Clinic Craving (From Pre-dose to Approximately 4-6 Hours Post-dose; and From Test Day 1 to Test Day 4 or 1 Week) - Via the Heroin Craving Questionnaire (HCQ)
Description: Subjects will be asked to complete the short version of the HCQ on their own time at home and bring it with them when they return for their next visit. Upon arrival to the clinic, subjects will also complete an HCQ with the coordinator to assess daily baseline cravings. This questionnaire will help us assess changes in craving generated outside of the clinical laboratory session from test day 1 through test day 4 (1 week later). Each item is scored on a scale ranging from 1 for "Strongly Disagree" to 7 for "Strongly Agree." Sum of all 14 items are scored and added. Mean scores reported below. Total Score Range: 14 (less cravings) - 98 (more cravings).
Time Frame: HCQ: once in clinic pre-dose at each test day, and once at home after each test day.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control | CBD 400mg | CBD 800mg
Number analyzed (Participants) | 15 | 14 | 13
units on a scale
  Session 1: Pre Drug/Placebo (Baseline) | 60.13 [56.36 to 63.91] | 59.33 [53.87 to 64.80] | 59.75 [54.72 to 64.78]
  Session 1: Post (At Home) | 53.20 [47.86 to 58.54] | 50.00 [43.23 to 56.77] | 53.42 [46.23 to 60.60]
  Session 2: Pre Drug/Placebo (Day 2 Baseline) | 53.40 [49.88 to 56.92] | 52.00 [45.33 to 58.67] | 51.17 [45.13 to 57.20]
  Session 2 Post (At Home) | 54.80 [49.70 to 59.90] | 49.47 [42.32 to 56.61] | 54.92 [45.50 to 64.33]
  Session 3: Pre Drug/Placebo (Day 3 Baseline) | 52.67 [46.84 to 58.49] | 50.87 [43.65 to 58.08] | 53.92 [45.79 to 62.04]
  Session 3 Post (At Home) | 52.21 [48.92 to 55.51] | 50.20 [43.79 to 56.61] | 55.40 [47.88 to 63.12]
  Session 4: Drug/Placebo (Day 4 Baseline) | 53.53 [50.11 to 56.95] | 49.67 [42.83 to 56.50] | 52.09 [41.81 to 62.37]

3. Secondary Outcome: Vital Signs
Description: Blood pressure (in mmHg), heart rate (in beats/min), temperature (in degrees Fahrenheit), respiratory rate (in breaths/min), and O2 saturation and pain will be monitored throughout the time course of the study and changes from baseline will be studied across the various time points. Note, cue sessions occur consecutively in the same test day.
  Results reported below are responses from baseline following exposure to neutral and heroin-associated cues in Session 1 in subjects with CBD or placebo administration.
Time Frame: Pre-placebo/drug, -60 min pre-cue, -40 min pre-cue, -20 min pre-cue, cue (time 0), 15 min post-cue, 35 min post-cue, 50 min post-cue, 65 min post-cue, 85 min post-cue
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Control | CBD 400mg | CBD 800mg
Number analyzed (Participants) | 15 | 14 | 13
beats per minute
  Session 1 baseline pre-neutral cue | 76.75 (11.889) | 76.30 (11.295) | 78.00 (10.970)
  Session 1 -60 min pre-neutral cue | 76.25 (10.899) | 75.80 (10.789) | 77.57 (10.390)
  Session 1 -40 min pre-neutral cue | 74.13 (13.943) | 76.10 (12.662) | 74.14 (10.270)
  Session 1 -20 min pre-neutral cue | 73.63 (13.223) | 75.10 (11.638) | 73.29 (9.844)
  Session 1 cue (time 0) pre-neutral cue | 73.75 (14.119) | 72.80 (12.874) | 74.43 (11.312)
  Session 1 15 min post-neutral cue | 71.63 (15.747) | 74.70 (11.136) | 73.57 (11.178)
  Session 1 35 min post-neutral cue | 71.00 (15.657) | 72.60 (10.511) | 71.43 (8.284)
  Session 1 50 min post-neutral cue | 70.25 (14.230) | 70.40 (9.755) | 68.57 (7.044)
  Session 1 65 min post-neutral cue | 69.38 (12.883) | 68.80 (8.954) | 66.71 (6.849)
  Session 1 85 min post-neutral cue | 68.75 (13.328) | 69.70 (10.935) | 71.14 (10.090)
  Session 1 baseline pre-drug cue | 76.83 (10.187) | 71.00 (12.166) | 74.40 (5.413)
  Session 1 -60 min pre-drug cue | 77.50 (11.005) | 71.40 (11.845) | 73.80 (6.535)
  Session 1 -40 min pre-drug cue | 76.50 (9.955) | 70.20 (9.935) | 68.80 (4.324)
  Session 1 -20 min pre-drug cue | 74.00 (9.445) | 72.00 (9.695) | 69.20 (4.764)
  Session 1 cue (time 0) pre-drug cue | 72.67 (10.013) | 70.00 (9.592) | 68.00 (4.359)
  Session 1 15 min post-drug cue | 74.50 (10.521) | 69.00 (8.718) | 67.20 (2.775)
  Session 1 35 min post-drug cue | 74.50 (11.879) | 66.80 (10.085) | 66.00 (3.391)
  Session 1 50 min post-drug cue | 77.33 (7.607) | 69.80 (10.569) | 67.40 (2.881)
  Session 1 65 min post-drug cue | 76.00 (10.770) | 66.40 (9.423) | 67.40 (2.881)
  Session 1 85 min post-drug cue | 73.67 (10.875) | 68.00 (7.842) | 65.20 (3.114)

4. Other Pre Specified Outcome: CBD Effects on Cognitive Behavior
Description: Digit Span Backwards (DSB) is a memory task consisting of a span of digits recalled in reverse order. Participants are read a series of digits (e.g., 4,7,1) and must immediately repeat them back in reverse order (e.g., 1,7,4). Mean correct response times (hits) are reported below in milliseconds. Shorter response times indicate better participant outcomes.
  Digit Symbol Substitution Task (DSST) is a neuropsychological test consisting of digit-symbol pairs.The goal is to complete as many correct patterns as possible in 3 mins. Mean response times reported below in ms, with shorter times indicating better outcomes.
Time Frame: 2 times: once at pre-screening and once at test day 4, within 2 weeks of each other.
Measure: Mean (Standard Deviation); unit: units on a scale (ms)
Arm/Group | Control | CBD 400mg | CBD 800mg
Number analyzed (Participants) | 15 | 14 | 13
units on a scale (ms)
  Digit Symbol Substitution Test (DSST) - Pre·Screen Response Time (ms) | 12.99 (5.2) | 11.68 (11.2) | 15.83 (27.0)
  Digit Symbol Substitution Test (DSST) - Test Day 4 Response Time (ms) | 11.81 (4.2) | 7.09 (5.1) | 8.73 (4.6)
  Digit-Span Backwards (DSB) - Pre·Screen Response Time (ms) | 79.48 (80.9) | 76.07 (37.4) | 71.6 (33.4)
  Digit-Span Backwards (DSB) - Test Day 4 Response Time (ms) | 93.35 (43.1) | 97.57 (59.6) | 92.27 (40.8)

5. Other Pre Specified Outcome: Visual Analog Scale for Anxiety (VASA)
Description: Questionnaires will be used to measure subjective responses. Anxiety will be assessed using a visual analog scale for anxiety (VASA). VASA scale ranges from 0 for "Not Anxious at All" to 10 for "Extremely Anxious." Note, cue sessions occur consecutively in the same test day.
Time Frame: Test day I, II and IV: on arrival, baseline for cue sessions 1 and 2, post-cue sessions I and 2 (30 min from baseline), prior to discharge (approximately 2.5 hours from test day start on average); Test day III: on arrival and prior to discharge.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | CBD 400mg | CBD 800mg
Number analyzed (Participants) | 15 | 14 | 13
score on a scale
  First Baseline (before cue video) Session 1 | 1.93 (1.751) | 2.86 (1.956) | 3.77 (2.833)
  First Baseline (before cue video) Session 2 | 1.40 (1.682) | 1.29 (1.541) | .85 (1.463)
  First Baseline (before cue video) Session 4 | .87 (1.246) | 1.29 (1.490) | 1.25 (2.006)
  First Post Cue Session 1 | 2.87 (2.924) | 3.21 (1.626) | 3.54 (2.989)
  First Post Cue Session 2 | 1.80 (1.897) | 2.07 (2.303) | 1.31 (2.016)
  First Post Cue Session 4 | 1.33 (1.915) | 1.50 (1.345) | 1.67 (2.498)
  Second Base Line (before cue video) Session 1 | 1.80 (2.178) | 1.64 (1.906) | 2.77 (2.803)
  Second Base Line (before cue video) Session 2 | 1.40 (1.352) | 1.64 (2.205) | .92 (1.382)
  Second Base Line (before cue video) Session 4 | .73 (1.223) | 1.86 (2.381) | 1.42 (2.065)
  Second Post Cue Session 1 | 2.13 (2.264) | 1.43 (1.910) | 1.54 (1.664)
  Second Post Cue Session 2 | 1.80 (2.178) | 2.29 (2.463) | 1.15 (1.772)
  Second Post Cue Session 4 | 1.13 (1.302) | 1.14 (1.875) | .75 (.965)
  Post Relaxation video Session 1 | .40 (.632) | 1.07 (1.269) | .92 (1.188)
  Post Relaxation video Session 2 | .93 (1.223) | 1.29 (1.590) | .46 (.967)
  Post Relaxation video Session 4 | .33 (1.047) | .71 (.994) | .50 (.798)

6. Other Pre Specified Outcome: The Positive and Negative Affect Schedule(PANAS)
Description: Questionnaires will be used to measure subjective responses. The Positive and Negative Affect Schedule will allow us to obtain positive and negative affect measures and observe their changes from baseline over the course of the cue-induced craving session. Note, cue sessions occur consecutively in the same test day. Positive affect scores range from 10 - 50. Higher scores represent higher levels of positive affect. Negative affect scores range from 10 - 50. Higher scores represent high levels of negative affect.
Time Frame: Baseline for cue sessions 1 and 2, post-cue sessions I and 2 (30 min from baseline) during test days I, II and IV.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | CBD 400mg | CBD 800mg
Number analyzed (Participants) | 15 | 14 | 13
score on a scale
  Session 1 Neutral Cue Positive PANAS | 1.48 (1.07) | -0.29 (0.92) | -0.92 (1.51)
  Session 1 Drug Cue Positive PANAS | -0.45 (1.23) | 2.7 (1.32) | -2.1 (1.3)
  Session 2 Neutral Cue Positive PANAS | -1.93 (1.79) | 1.64 (0.99) | 0.26 (0.82)
  Session 2 Drug Cue Positive PANAS | 0.71 (0.64) | 1.08 (1.4) | -2.37 (1.52)
  Session 3 Neutral Cue Positive PANAS | 0.58 (0.78) | 2.21 (0.83) | 2.79 (1.15)
  Session 3 Drug Cue Positive PANAS | 1.52 (0.85) | 0.43 (1.26) | 4.05 (1.36)
  Session 1 Neutral Cue Negative PANAS | -0.51 (0.83) | -0.69 (0.97) | -1.48 (1.22)
  Session 1 Drug Cue Negative PANAS | 5.31 (1.85) | 1.26 (1.93) | 0.7 (1.33)
  Session 2 Neutral Cue Negative PANAS | -3.75 (0.79) | -3.01 (0.88) | -2.68 (1.03)
  Session 2 Drug Cue Negative PANAS | 1.18 (1.62) | 1.12 (1.81) | 1.76 (1.34)
  Session 3 Neutral Cue Negative PANAS | -0.06 (0.52) | -0.98 (0.74) | -0.14 (0.5)
  Session 3 Drug Cue Negative PANAS | 1.32 (0.9) | 0.77 (0.71) | 0.57 (0.74)

7. Other Pre Specified Outcome: Physiological Response to Stress - Salivary Cortisol Measures
Description: Subjects will be asked to chew on a cotton swab, each time providing us with a saliva sample from which we can detect free cortisol levels and extrapolate serum levels of the stress indicator affected by the video cues. Note, cue sessions occur consecutively in the same test day. Thus, the physiological stress of craving will be monitored and measured across the multiple time points to observe any changes from baseline.
  Results reported below are mean percent change from baseline following exposure to neutral and heroin-associated cues in Session 1 in subjects with CBD or placebo administration.
Time Frame: Test day I: 15 min and 35 min post drug and neutral cue
Measure: Mean (Standard Error); unit: mean percent change
Arm/Group | Control | CBD 400mg | CBD 800mg
Number analyzed (Participants) | 15 | 14 | 13
mean percent change
  Neutral Cue 15 min | 0.69 (3.45) | 1.19 (6.19) | -0.87 (4.11)
  Neutral Cue 35 min | -3.84 (6.00) | -9.82 (5.93) | -4.17 (7.15)
  Drug Cue 15 min | 11.89 (6.70) | -15.17 (7.42) | -13.84 (11.70)
  Drug Cue 35 min | 8.19 (10.98) | -23.74 (6.66) | -20.03 (8.54)

8. Other Pre Specified Outcome: Adverse Effects - SAFTEE
Description: Before being sent home, subjects will be asked to complete the Systematic Assessment for Treatment of Emergent Events (SAFTEE) to ensure that they are not experiencing any negative effects of the treatment. There will also be a debriefing period at the end of each session aimed to minimize any potential increase in craving beyond the clinical laboratory session. At the end of the last study, subjects will be assessed and offered appropriate resources and guidance for seeking help for substance abuse or cravings should they need it after participation in the study has concluded.
Time Frame: Test day I, II, III and IV: at the end of day prior to discharge. Average time point: approximately 150 minutes into the test day.
Measure: Number; unit: events
Arm/Group | Control | CBD 400mg | CBD 800mg
Number analyzed (Participants) | 15 | 14 | 13
events
  Headache | 2 | 1 | 0
  Joint Pain | 1 | 0 | 0
  Tired/Fatigue | 2 | 0 | 1
  Chest Pain | 0 | 1 | 0
  Eye Irritation | 0 | 1 | 0
  Abdominal Discomfort | 0 | 0 | 1
  Diarrhea | 0 | 2 | 7

9. Other Pre Specified Outcome: CBD Effects on Cognitive Behavior
Description: Continuous Performance Test is a computerized assessment of attention. The outcome measures include correct responses (hits), missed responses (misses), incorrect responses (false hits), correct misses, and reaction time of both hits and misses. Mean correct response times (hits) are reported below. Shorter response times indicate better participant outcomes.
Time Frame: 2 times: once at pre-screening and once at test day 4, within 2 weeks of each other.
Measure: Mean (Standard Deviation); unit: units on a scale (hits)
Arm/Group | Control | CBD 400mg | CBD 800mg
Number analyzed (Participants) | 15 | 14 | 13
units on a scale (hits)
  Continuous Performance Task (CPT) - Pre-Screen Correct Responses (hits) | 40.73 (29.6) | 39.13 (17.2) | 40.67 (17.2)
  Continuous Performance Task (CPT) - Test Day 4 Correct Responses (hits) | 49.93 (12.1) | 46.2 (13.8) | 47.5 (14.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the course of study participation, approx. 2 weeks.
Description: Adverse events were collected by using SAFTEE (Systematic Assessment for Treatment Emergent Events)
Arm/Group | Control | CBD 400mg | CBD 800mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 3/15 | 4/14 | 5/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=15) | CBD 400mg (N=14) | CBD 800mg (N=13)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tired/Fatigue (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02539823/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02539823/SAP_001.pdf